CLINICAL TRIAL: NCT00801086
Title: Phase II Double-Blind, Placebo-Controlled Study of the Safety and Preliminary Effectiveness of MTS-01 for the Prevention of Alopecia Induced by Whole Brain Radiotherapy
Brief Title: Efficacy Study of Tempol to Prevent Hair Loss From Radiotherapy to the Brain
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mitos Pharmaceuticals (Industry)
Responsible Party: Louis Habash/ President and CEO, Mitos Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MITO 02-03
Record Dates: First submitted 2008-12-01; First posted 2008-12-03 (Estimated); Last update posted 2008-12-03 (Estimated); Status verified 2008-12

CONDITIONS: Alopecia
Keywords: Alopecia; Hair loss; Radiation; Whole brain radiotherapy; Radiation-induced alopecia
MeSH Terms: conditions — Alopecia | interventions — tempol; Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): MTS-01 (7% Tempol gel)
  Interventions: Drug: 7% (w/v) Tempol alcohol-based gel (MTS-01)
- 2 (Placebo Comparator): Vehicle
  Interventions: Drug: alcohol-based gel

INTERVENTIONS:
Drug: 7% (w/v) Tempol alcohol-based gel (MTS-01) — 200mL gel applied daily prior to radiation dose and removed immediately thereafter.
  Arms: 1
Drug: alcohol-based gel — 200mL gel applied daily prior to radiation dose and removed immediately thereafter
  Arms: 2

SUMMARY:
Hair loss occurs commonly as a result of radiotherapy administered to the brain, and this can contribute to the distress and social isolation of patients with advanced cancer. In this study a topical gel will be applied directly to the scalp during each dose of radiotherapy. The goal is to determine to what extent the experimental drug is successful in lessening the hair loss.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic cancer to the brain for which palliative whole brain radiotherapy is recommended.
* Hair that covers the scalp and is at least 1/4 inch in length

Exclusion Criteria:

* Receiving chemotherapy known to cause alopecia within 60 days of study or during the study.
* Pre-existing alopecia
* Previous brain radiotherapy
* scalp metastases or scalp wounds
* use of hair dyes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-12 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Effectiveness will be based on a comparison of hair retention scores between MTS-01 and placebo. | Assessments occur weekly during treatment and follow-up assessments occur for 12 weeks following treatment.

CONTACTS AND LOCATIONS:
Overall Officials: James Metz, MD, Study Chair — University of Pennsylvania
Locations (2):
- United States (2):
  - University of Arizona, Tucson, Arizona
  - University of Pennsylvania, Philadelphia, Pennsylvania